CLINICAL TRIAL: NCT00558454
Title: Randomized, Controlled Study of Iron Supplementation of Infants With Birth Weights 2000-2500 g
Brief Title: Iron Supplementation of Marginally Low Birth Weight Infants
Acronym: JOHN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Jerring Foundation, Sweden (Unknown); Oskar Foundation (Other)
Responsible Party: Principal Investigator, Magnus Domellöf, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Iron for LBW infants
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Anemia; Iron-Deficiency; Child Behavior Disorders; Cognitive Manifestations
Keywords: Iron supplements; Infant; Low birth weight; Prevention of iron deficiency and its physiological consequences; Safety
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Child Behavior Disorders; Neurobehavioral Manifestations | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Iron
- 2 (Experimental): 1 mg/kg/day from age 6 weeks to 6 months
  Interventions: Drug: Iron
- 3 (Experimental): 2 mg/kg/day from age 6 weeks to 6 months
  Interventions: Drug: Iron

INTERVENTIONS:
Drug: Iron — Ferrous succinate mixture
  Other Names: Ferromyn S, AstraZeneca, Södertälje, Sweden

SUMMARY:
Iron is essential for brain development and there is a well established association between iron deficiency in infants and poor neurological development. In Sweden, about 5% of newborns have low birth weight (< 2500 g). Due to small iron stores at birth and rapid postnatal growth, they have increased risk of iron deficiency and it is therefore important to prevent iron deficiency in this population. However, excessive iron supplementation can have adverse effects in infants such as growth impairment. In a randomized, controlled trial, we are investigating the effects of 0, 1 or 2 mg/kg/d of iron on brain myelination, cognitive development and growth in low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Marginally low birth weight (2000-2500 g)
* Healthy at inclusion(6 weeks of age)
* No previous blood transfusion
* No previous iron supplementation

Exclusion Criteria:

* Anemia at inclusion

Ages: 39 Days to 45 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Neurological developement | 6 months, 3 years and 7 years
  6 mo: Auditory brain stem response (central conduction time) 3 y: CBCL - Parental questionnaire assessing behavioral problems and WIPPSI - test of cognitive functions 7 y: SDQ, 5-15 and CBCL - Parental questionnaires assessing behavioral problems, TeAch - test of behavioral problems and WISC - test of cognitive functions.

SECONDARY OUTCOMES:
Growth (weight, length, head circumference, knee-heel length), Morbidity and Iron status (Hemoglobin, ferritin etc) | 6 months
Growth, Iron status, and Morbidity | 3 years and 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Domellöf, MD, PhD, Principal Investigator — Umeå University, Sweden
Locations (2):
- Sweden (2):
  - Karolinska Hospital (including Danderyd Hospital), Stockholm
  - Umeå University Hospital, Umeå

REFERENCES:
- [Derived] Lindberg J, Norman M, Westrup B, Domellof M, Berglund SK. Lower systolic blood pressure at age 7 y in low-birth-weight children who received iron supplements in infancy: results from a randomized controlled trial. Am J Clin Nutr. 2017 Aug;106(2):475-480. doi: 10.3945/ajcn.116.150482. Epub 2017 Jun 28. PMID 28659293
- [Derived] Lindberg J, Norman M, Westrup B, Ohrman T, Domellof M, Berglund SK. Overweight, Obesity, and Body Composition in 3.5- and 7-Year-Old Swedish Children Born with Marginally Low Birth Weight. J Pediatr. 2015 Dec;167(6):1246-52.e3. doi: 10.1016/j.jpeds.2015.08.045. Epub 2015 Sep 26. PMID 26394823
- [Derived] Berglund SK, Westrup B, Domellof M. Iron supplementation until 6 months protects marginally low-birth-weight infants from iron deficiency during their first year of life. J Pediatr Gastroenterol Nutr. 2015 Mar;60(3):390-5. doi: 10.1097/MPG.0000000000000633. PMID 25406528
- [Derived] Berglund SK, Lindberg J, Westrup B, Domellof M. Effects of iron supplements and perinatal factors on fetal hemoglobin disappearance in LBW infants. Pediatr Res. 2014 Nov;76(5):477-82. doi: 10.1038/pr.2014.116. Epub 2014 Aug 13. PMID 25119339
- [Derived] Berglund SK, Westrup B, Hagglof B, Hernell O, Domellof M. Effects of iron supplementation of LBW infants on cognition and behavior at 3 years. Pediatrics. 2013 Jan;131(1):47-55. doi: 10.1542/peds.2012-0989. Epub 2012 Dec 10. PMID 23230066
- [Derived] Berglund S, Lonnerdal B, Westrup B, Domellof M. Effects of iron supplementation on serum hepcidin and serum erythropoietin in low-birth-weight infants. Am J Clin Nutr. 2011 Dec;94(6):1553-61. doi: 10.3945/ajcn.111.013938. Epub 2011 Nov 9. PMID 22071701
- [Derived] Berglund S, Westrup B, Domellof M. Iron supplements reduce the risk of iron deficiency anemia in marginally low birth weight infants. Pediatrics. 2010 Oct;126(4):e874-83. doi: 10.1542/peds.2009-3624. Epub 2010 Sep 6. PMID 20819898